CLINICAL TRIAL: NCT02865902
Title: Low-level Laser Therapy in Enhancing Wound Healing and Preserving Tissue Thickness at Free Gingival Graft Donor Sites: A Randomised Controlled Clinical Study
Brief Title: Low-level Laser Therapy in Enhancing Wound Healing and Preserving Tissue Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Gülbahar Ustaoğlu, Reseach Asistant, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24237859-545
Record Dates: First submitted 2016-08-01; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Wounds
Keywords: Low level laser therapy; wound healing; periodontology
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Experimental): In Test group, the free gingival graft donor sites of each experimental group received low-level laser therapy by Ezlase; Biolase® at doses of 8.6 J/cm2.
  Interventions: Device: Low-Level Laser Therapy by Ezlase; Biolase®
- Control Group (Sham Comparator): In Control Group, the low-level laser therapy by Ezlase; Biolase® was performedin a same manner with test group at free gingival graft donor sites. However, no irradiation was occurred because of not pushing the start button.
  Interventions: Device: Low-Level Laser Therapy by Ezlase; Biolase®

INTERVENTIONS:
Device: Low-Level Laser Therapy by Ezlase; Biolase® — comparision of the effects of low-level-laser therapy on wound healing of palatal donor site

SUMMARY:
Objective: The aim of this study was to determine the effects of Low Level Laser Therapy (LLLT) on wound healing at Free Gingival Graft donor sites (FGGDS).

Materials and Methods: Forty patients requiring FGG were selected for this randomized controlled double blinded prospective clinical trial. The FGGDS were treated with LLLT and compared with an untreated control group. The Wound Healing Index (WHI), tissue consistency, colour match (CM), and H2O2 bubbling test for the evaluation of complete wound epithelialization (CWE) were recorded at the 3rd, 7th, 14th and 21st days. The pain-burning level, number of analgesics, and bleeding were recorded for 7 days. Donor area soft tissue thickness (TT) was measured at baseline and at the 1st month.

DETAILED DESCRIPTION:
Subjects and Study Design This single center, randomized, double blinded, prospective and controlled clinical study was performed to evaluate the healing time, wound epithelialization and post-operative morbidity produced after harvesting FGG from the palate. The wounds were treated with one of the following methods: sterile wet gauze pressure (control) or LLLT (test).

The patients were randomly assigned to one of the groups by the periodontists with the toss of a coin.

Forty patients requiring FGG were selected, and verbal and written informed consent were obtained.

To minimize the differences related to the surgical technique, all surgical procedures were carried out by one experienced clinician.

Pre-Surgical Treatments All selected patients underwent a professional periodontal prophylaxis phase, and all patients were given proper oral hygiene instructions. Patients who had a full mouth plaque score (FMPS)˂20% and a full mouth bleeding score (FMBS)˂20% were included in the study. The patients were assigned to the control or test groups by the coin toss method.

Surgical Procedure After local anaesthesia, the free gingival graft was harvested as follows: the donor site extended from the distal line angle of the canine to the mesial line angle of the maxillary first molar by conventional scalpel. An approximately 1.5 mm split-thickness and rectangular-shaped (7x12 mm) gingival graft was obtained. The free gingival graft was sutured to the prepared recipient bed using size 5-0 resorbable sutures.

Test Group - LLLT The Ga-Al-As laser was used for LLLT at a wavelength of 940 nm. The wounds of each experimental group received laser stimulation at doses of 8.6 J/cm2, very closed the described dose (10 J/cm2) in the literature. The power output was maintained at a constant 3 W in the continuous-wave (cw) mode; the pulse interval size was 0.10 ms, and the pulse length was 0.05 ms. Laser energy was applied via a 400-µm optical fibre with a Whitening and Pain Relief Handpiece® . The handpiece was positioned at a distance of approximately 1 mm proximal to the wound area perpendicularly at a non-contact mode. The spot area of handpiece involved all the wound area . The application area was actually similar with the probe spot area (2.8 cm2). The wound area was 7x12=0.84 cm2. So the spot area of the probe was wider than the wound area and included all the wound area. For this reason, we did not need to move the handpiece, only kept constant. All surfaces of the wound were irradiated leading to total dosage of 8.6 J/cm2 and the irradiation time was 8 s. The energy at the wound area was 7.2 J (0.84 cm2 x 8.6 J/cm2 =7.2 J). The specified laser dose was initiated after surgery and was repeated on the 3rd, 5th, and 7th days after operation. The cumulative dose was 34.4 J/cm2 at total.

Control Group - LLLT Sham Sterile wet gauze was pressed to the FGG donor site for 5 min in the control group. The LLLT was performed in a same manner with test group. However, no irradiation was occurred because of not pushing the start button.

Post operative care A non-eugenol pack was placed over the sutured FGG (Coe-Pak™ Periodontal Dressing, GC America Inc., IL, USA). An acrylic stent was prepared to protect the palatal donor site and placed after surgery and recommended to patients to wear for 7 days. Patients were prescribed 500 mg of paracetamol (if needed) and a 0.12% chlorhexidine oral rinse twice a day for 2 weeks. The patients were advised to report any adverse outcomes and were recalled at 3rd, 7th, 14th, 21st and 30th day (the 5th day for the LLT group). The sutures were removed after 2 weeks.

Evaluated Parameters All evaluations were acquired by one periodontist who was blinded to the treatment assignment. The following parameters were recorded: H2O2 bubbling test for screening complete epithelialization, the Landry Wound Healing Index (WHI), pain and burning sensations by a VAS score, bleeding (yes/no), palatal tissue consistency, colour match, tissue thickness, and the number of analgesics.

Intra-Surgical Measurements of Soft Tissue Thickness The thickness of the palatal soft tissue in the harvesting area was measured after local anaesthesia. The measurement was made approximately 5 mm apical to the gingival margin of the first premolar by means of a #20 endodontic reamer with a silicon stopper. The thickness of the palatinae was measured in the test and control groups. The penetration depth was measured with a digital caliper. The dimensions of the graft were standardized by a sterile aluminium foil template that was 7x12 mm in dimension.

Subjective Assessments During the 7 days after the FGG procedure, the patients were asked to keep a diary of pain and burning sensations using a Visual Analogue Scale (VAS) to evaluate the intensity of the given event. The VAS score for pain ranged from 0 (no pain) to 100 (severe pain), represented by a continuous line of 10 cm length; while the burning sensation was scored as follows: 0 (absent) to 100 (severe burning). Additionally, the patients were asked to report their postoperative bleeding for 7 days as "Bleeding present (+)" or "Bleeding absent (-)".

Palatal Tissue Consistency The consistency of the palatal mucosa was assessed on the 3rd, 7th, 14th and 21st days by palpation with a blunt instrument and was scored as soft or firm by a clinician who was blind to the treatment assignment.

Colour match On the 3rd, 7th, 14th and 21st days, the colour of the palatal mucosa was assessed by comparing it to that of the adjacent and opposite side using the objective VAS (VAS score 0-100) represented by a continuous line of 10 cm length, by a clinician blinded to the treatment group assignment. A score of 0 indicated no colour match, and a score of 100 indicated a very good colour match with the adjacent tissues.

Wound Epithelialization CWE (complete Wound Epithelialization) was evaluated clinically by the peroxide bubbling test . This was the primary outcome of this study. This test is based on the principle that if the epithelium is discontinuous, then H2O2 diffuses into the connective tissue, and the enzyme catalase acts on H2O2 to release water and oxygen, which is clinically observed as the production of bubbles on the wound. The area to be evaluated was dried, and 3% H2O2 was sprinkled on the wound with a syringe, followed by a period of waiting (approximately 10 seconds) for the appearance of bubbles, which suggest that the surgical site was not completely epithelialized.

Landry Wound Healing Index (WHI) The palatal wounds were scored using the Landy Wound Healing Index on the 3rd, 7th, 14th and 21st days post operatively. This index evaluated the wounds based on the following criteria: tissue colour, response to palpation, incision margins and suppuration. The scores range from 1-5 and correspond to very bad to excellent healing.

The number of analgesics Patients were asked to record the number of analgesics taken for pain relief during the first 7 post-operative days.

Statistical Analysis The homogeneity of the data was tested by the Shapiro Wilk test. Non-parametric tests were used. SPSS v.17.0 (SPSS Inc., Chicago, Illinois USA) was used for the analysis. The Mann-Whitney U test was used to analyze intergroup differences. Time dependent alterations were analyzed by the Wilcoxon test. The Binary Logistic Regression Analysis was performed to analyze the factors that affect epithelialization. Significance level was p<0.05.

Power Calculation The primary outcomeof this study were the H2O2 test results. The power analysis was performed with ttp://www.openepi.com/Menu/OE_Menu.htm. The power of this study was calculated as 98.86%.

ELIGIBILITY:
Inclusion Criteria:

1. The absence of systemic factors (no systemic disease, no coagulation disorders, no medications affecting periodontal status, and no pregnancy or lactation)
2. No smoking
3. Patients who had a full mouth plaque score (FMPS)˂20% and a full mouth bleeding score (FMBS)˂20%
4. No periodontal surgery on the experimental site
5. No nauseal reflection

Exclusion Criteria:

1. Smoking
2. The presence of systemic disease
3. Bad oral hygiene-
4. The history of periodontal surgery on the experimental site
5. Nauseal reflection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Complete Wound Epithelization | 14th. day after surgery
  The 14th day H2O2 Bubbling test results that show Complete Wound Epithelization

SECONDARY OUTCOMES:
Palatal Tissue Thickness | at baseline and at the 1st month
  The tissue thickness alterations (mm.) that was measured by a endodontic reamer and digital caliper was the secondary outcome

IPD SHARING:
Plan to Share IPD: Undecided